CLINICAL TRIAL: NCT03681392
Title: A Phase 2 Open-label Randomized Crossover Dose-finding Study of the Efficacy, Safety, and Tolerability of Dr. Pyke's Supplement for Stream (S4S) in Older Men With Lower Urinary Tract Symptoms and/or Sexual Dysfunction
Brief Title: Study of Dr. Pyke's Supplement for Stream (S4S) in Men With Prostatism and ED
Acronym: S4S4BPH/ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Robert E. Pyke (Industry)
Responsible Party: Sponsor-Investigator, Robert E. Pyke, Trial Investigator, drpykessupplements.com
Organization: drpykessupplements.com (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pykonsult 2001
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Prostatism; Erectile Dysfunction
Keywords: Benign Prostatic Hypertrophy; Erectile Dysfunction; Nutritional Supplements; Prostatism; Lower Urinary Tract Symptoms, male
MeSH Terms: conditions — Prostatism; Erectile Dysfunction; Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Rivers

STUDY DESIGN:
Intervention Model Description: Randomized open-label crossover design with 1:1 allocation of first regimen as once daily or twice daily
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Once daily then twice daily (Experimental): One 6.5 cc scoop of S4S once a day for 7 days, then one 6.5 cc scoop of S4S twice a day for 7 days
  Interventions: Dietary Supplement: Dr. Pyke's Supplement for Stream (S4S)
- Twice daily then once daily (Experimental): One 6.5 cc scoop of S4S twice a day for 7 days, then one 6.5 cc scoop of S4S once a day for 7 days
  Interventions: Dietary Supplement: Dr. Pyke's Supplement for Stream (S4S)

INTERVENTIONS:
Dietary Supplement: Dr. Pyke's Supplement for Stream (S4S) — Proprietary combination of Panax ginseng extract, L-citrulline, beta-sitosterol and vitamin D3
  Other Names: S4S

SUMMARY:
This is the first clinical trial of Dr. Pyke's Supplement for Stream (S4S), a proprietary combination of Panax ginseng extract, L-citrulline, beta-sitosterol and vitamin D3, to investigate its effects on prostatism and erections, and its tolerability, when taken daily and twice-daily for 2 weeks.

DETAILED DESCRIPTION:
This is a 2-week clinical trial of Dr. Pyke's Supplement for Stream (S4S), a proprietary combination of Panax ginseng extract, L-citrullline, beta-sitosterol and vitamin D3, investigating its lower urinary tract effects, sexual effects, and tolerability in two dose regimens-daily for a week and twice daily for a week--in men who have Lower Urinary Tract Symptoms (LUTS) and may have erectile dysfunction (ED). No clinic visits are required. Subjects will be consented, screened, supplied with S4S, and tested via the Internet. Subset analyses will evaluate effects in three populations: men with at least moderate lower urinary tract symptoms (LUTS), according to standard score cutoff; men with at least moderate Erectile Dysfunction (ED, according to standard score cutoff; and all men dissatisfied with their urinary function and meeting minimal criteria for inclusion.

ELIGIBILITY:
Inclusion Criteria:

Inclusion requirements for all subjects

1. Men at least 40 years of age
2. Screening IPSS QoL must be 4-6:

   If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Delighted (0), Pleased (1), Mostly Satisfied (2), Mixed (3), Mostly Dissatisfied (4), Unhappy (5), Terrible (6)
3. Gives informed consent for study and is willing to take the treatments and complete the scheduled evaluations
4. Willing to buy S4S for $30, with the understanding that a rebate of $30 or a coupon for $30 off the cost of a second 30-dose supply of S4S will be offered if the subject completes the electronic questionnaires at the end of the treatment

Required for target efficacy subset

Meets criterion for at least moderate ED: IIEF-5 (erectile function) score <13 - or:

Meets criterion for at least moderate Lower urinary tract symptoms (LUTS): IPSS score at least 20

Exclusion Criteria:

1. Known allergy or sensitivity to ginseng, L-citrulline, canola oil or soybean oil.
2. Current severe side effects from any drug
3. Using medication(s) for angina pectoris, LUTS, or ED and has not consulted personal physician on advisability of participating in this study.
4. Women

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male prostate gland dysfunction is required
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score (IPSS) | 1-4 weeks
  measure of lower urinary tract symptoms in men with prostatism, total score; 0=best possible (no symptoms); 35 = worst possible; mean change and number of patients 50% improved
Primary safety outcome: adverse events | 1 week
  Reports from subjects of new or worse symptoms; number of patients with any adverse event, count and % of patients with each type of such adverse events

SECONDARY OUTCOMES:
Secondary safety outcome: Adverse event dropouts | 1-2 weeks
  Reports from subjects; number and % of patients
International Prostate Symptoms Scale Quality of Life due to urinary symptoms | 1-4 weeks
  categorical single-item self-report from "delighted" to "terrible" plus brief write-in; % improving by at least 1 point
Volunteer's Global Impression of Change in Erectile function | 1 week
  categorical single-item self-report from "very much improved" to "worse" plus brief write-in; % improvement by at least 1 point
International Index of Erectile Function (IIEF)-5 | 1-4 weeks
  5-item cluster on erectile function, score = 5 (worst possible) to 25 (completely normal); mean change and % improving by at least 2 points

OTHER OUTCOMES:
Serious adverse events | 2 weeks
  Rate of reported diagnoses from treating physicians if any subjects are hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Pyke, MD, PhD, Study Director — Pykonsult LLC

IPD SHARING:
Plan to Share IPD: Undecided
Yes

REFERENCES:
- [Background] Pyke RE. Exo-Clinical Trials of Nutritional Supplements for Sexual Dysfunction: Precedents, Principles, and Protocols. Sex Med Rev. 2019 Apr;7(2):251-258. doi: 10.1016/j.sxmr.2018.07.002. Epub 2018 Oct 6. PMID 30301704